CLINICAL TRIAL: NCT07016542
Title: Cohort for Monitoring Patients With Venous Thromboembolic Disease
Acronym: CoMTEV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/352/OB; ID RCB : 2018-A02844-51 (Other: ANSM)
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Venous Thromboembolic Disease
Keywords: risk of thrombotic recurrence; hemorrhagic risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient having experienced at least one venous thromboembolic episode

SUMMARY:
Venous thromboembolic disease is a common pathology in the general population (1.5/1000), the prognosis of which depends in particular on the risk of recurrence. This risk depends essentially on whether the thrombotic episode was provoked or not. Thus, patients who present a thromboembolic event without any contributing factor have a high risk of recurrence, which encourages clinicians to continue anticoagulant treatment for a long time. However, anticoagulant treatment is the leading cause of hospitalization for iatrogenic causes and the leading cause of iatrogenic mortality. The benefit-risk balance of treatment must be evaluated regularly, which requires a good knowledge of the risk factors for thrombotic recurrence and the risk factors for hemorrhage.

DETAILED DESCRIPTION:
Several tools have been established and validated to help clinicians assess patients' bleeding risk, notably using the HAS BLED, haemorrage, and more recently the VTE BLED score. This latest score, published very recently, is the only one to have been validated in patients treated with direct oral anticoagulants. At the same time, we have recurrence risk scores such as HERDOO2, which allow us to identify patients at low risk of recurrence.

In order to improve the management of patients with venous thromboembolic disease, multidisciplinary thrombosis RCPs have been established since 2015, bringing together hemostasis specialists, internists, oncologists, and private vascular physicians to assist clinicians in managing complex cases. • Dedicated post-emergency consultations twice a week to streamline outpatient care for less serious patients This study aims to evaluate the effectiveness of these tools: score and RCP in the management of patients with venous thromboembolic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient over 18 years of age who has experienced at least one venous thromboembolic episode:

   * Deep vein thrombosis confirmed by Doppler ultrasound or CT venography,
   * Pulmonary embolism confirmed by CT angiography, ventilation/perfusion scan, or confirmed DVT episode with respiratory signs consistent with PE.
2. Hospitalization in the Internal Medicine Department
3. Consultation by an Internal Medicine physician
4. File presented at the thrombosis multidisciplinary meeting

Exclusion Criteria:

Thrombosis not meeting the inclusion criteria (cerebral venous thrombosis, mesenteric)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having experienced at least one venous thromboembolic episode
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2031-12-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence in patients treated with venous thromboembolic disease (VTE) | 12 years
  Evaluation of the number of hospitalizations or consultations for a venous thrombotic recurrence
Rate of bleeding complications in patients treated with venous thromboembolic disease (VTE) | 12 years
  Evaluation of the number of hospitalizations or consultations for a hemorrhagic complication.

SECONDARY OUTCOMES:
Long-term complication rates | At enrollment visit, 6 months, 1 years and each year during 12 years
  Assessment of the occurrence of long-term complications
Long-term complication rates | At enrollment visit, 6 months, 1 years and each year during 12 years
  Assessment of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien SM MIRANDA, Doctor, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
The data provided will be the property of the sponsor and will be used solely for its own research activities.
Supporting Information: SAP